CLINICAL TRIAL: NCT05420012
Title: The Effect of Vericiguat on Peripheral Vascular Function, Patient Health Status and Inflammation in Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: The Effect of Vericiguat on Peripheral Vascular Function, Patient Health Status and Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Josef Stehlik (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Josef Stehlik, Professor, Division of Cardiovascular Medicine, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00152530
Record Dates: First submitted 2022-06-11; First posted 2022-06-15 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction (HFrEF)
MeSH Terms: conditions — Heart Failure | interventions — vericiguat; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized double-blind, placebo-controlled study in patients with heart failure [HF] with reduced ejection fraction [HFrEF].
Who Masked: Participant, Investigator
Masking Description: Patients will be assigned with equal allocation to the intervention and control groups using block randomization to ensure a balance in sample size across groups over time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vericiguat (Experimental): Study drug
  Interventions: Drug: Vericiguat
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vericiguat — A starting dose of vericiguat 2.5 mg or matching placebo will be initiated after randomization and completion of the baseline testing. Subjects will be up-titrated in a blinded fashion to 5 mg and then to the target dose of 10 mg of vericiguat or matching placebo using titration criteria based on mean systolic blood pressure(SBP) evaluation and clinical symptoms at 2 week intervals. Titration to 10 mg in subjects who have not yet reached the target dose is intended at every visit/phone call throughout the study duration based on mean SBP measurement and safety considerations, at the discretion of the investigator.
  Other Names: VERQUVO
  Arms: Vericiguat
Drug: Placebo — A starting dose of vericiguat 2.5 mg or matching placebo will be initiated after randomization and completion of the baseline testing. Subjects will be up-titrated in a blinded fashion to 5 mg and then to the target dose of 10 mg of vericiguat or matching placebo using titration criteria based on mean systolic blood pressure(SBP) evaluation and clinical symptoms at 2 week intervals. Titration to 10 mg in subjects who have not yet reached the target dose is intended at every visit/phone call throughout the study duration based on mean SBP measurement and safety considerations, at the discretion of the investigator.
  Other Names: Control group
  Arms: Placebo

SUMMARY:
The concept that direct stimulation of soluble guanylate cyclase (sGC) could be a particularly effective approach to increase cyclic guanosine monophosphate (cGMP) in conditions of increased inflammation/oxidative stress, endothelial dysfunction, and reduced nitric oxide (NO) bioavailability. Thus, the aim of the proposed study is to examine the effect of Vericiguat on peripheral vascular function, inflammatory status, and patient health status. The study also aims to identify patients who are particularly likely to benefit from Vericiguat treatment and predict that these patients will be defined by baseline peripheral vascular dysfunction and high inflammatory state.

DETAILED DESCRIPTION:
The incidence of heart failure (HF) continues to increase, along with its associated morbidity, mortality, and cost. Novel therapeutic options have been proposed to address the needs of especially the patients who remain symptomatic despite optimal medical therapy. A number of factors lead to ongoing symptoms in patients with chronic heart failure (HF), including persistent abnormalities in myocardial function, neurohormonal dysregulation, and of the peripheral vascular system.

The Phase 3 VICTORIA trial examined the efficacy of Vericiguat, a novel oral soluble guanylate cyclase (sGC) stimulator in patients with HF and reduced ejection fraction (HFrEF). Vericiguat enhances the cyclic guanosine monophosphate (GMP) pathway by directly stimulating soluble guanylate cyclase independent of nitric oxide (NO). The VICTORIA study showed that patients who received Vericiguat 2.5 mg once daily up-titrated to 10 mg daily had a lower incidence of the primary endpoint of cardiovascular death or first HF hospitalization compared to placebo 1.

Determining the exact mechanism, or the respective contribution of different mechanisms, through which Vericiguat improves outcomes in HFrEF may allow for better tailoring of its use to individual patients. The preliminary results of an echocardiography sub-study indicate that there was no significant difference in the change of left ventricular ejection fraction (LVEF) between baseline and study end among patients assigned to the active drug vs placebo. We hypothesize that the beneficial effects of Vericiguat in HF may not be linked to improvement in myocardial contractility, but rather to the effects of sGC stimulation on the peripheral vasculature. This was not directly tested in VICTORIA.

Studies from our group 2, 3 and others 4, 5 have collectively identified a marked reduction in vascular function, as determined by flow-mediated vasodilation (FMD) testing, in patients with HFrEF despite optimized pharmacotherapy, indicative of a pervasive, disease-related reduction in endothelial health. Endothelial dysfunction is characterized by NO dysregulation, inflammation, and oxidative stress. These factors impair the capacity of the vascular endothelium to perform its numerous functions including regulation of vascular tone and inflammatory processes. Importantly, endothelial dysfunction is also associated with reduced quality of life 6 and decreased physical capacity 7, 8 in patients with HFrEF. These studies suggest that the consequences of vascular dysfunction are far-reaching and support the concept that interventions targeting the peripheral vasculature to induce systemic effects could prove beneficial in cardiovascular disease. This is particularly relevant given the known relationship between endothelial dysfunction and mortality risk in patients with HFrEF 9, 10. Improvement in peripheral vascular function in patients with HFrEF would in turn lead to improved physical capacity and health-related quality of life (hrQOL).

Preclinical studies provide evidence of sGC stimulation favorably affecting peripheral vascular function. In a rat model of HF, treatment with Ataciguat normalized endothelial function, improved sensitivity to NO, and reduced platelet activation 11. However, the impact of Vericiguat on vascular health has not been evaluated in human HF. A recent study also examined the effect of Vericiguat on inflammation and oxidative stress in HF 12. After 12 weeks of Vericiguat therapy, high sensitivity CRP (hsCRP) decreased significantly, and the probability of hsCRP value being ≤3.0 mg/L at the end of the study was higher in patients treated with Vericiguat compared to placebo. Although the impact of Vericiguat on upstream, inflammatory cytokines such as IL-1β and IL-18 have not been determined, there is strong evidence supporting elevation of these biomarkers that reflect NRLP3 inflammasome activation in patients with HFrEF13, 14. Given the recent success in clinical trials targeting the inflammasome in heart failure 15 and recent evidence for the efficacy of sGC stimulation to mitigate NLRP3 inflammasome activity in other organ systems 16, there is strong rationale for the expectation that Vericiguat may favorably impact both upstream (IL-1β, IL-18, TNF-α and IL-6) and downstream (hsCRP) inflammatory biomarkers. Importantly, an inverse correlation between biomarkers of inflammation and endothelial function has been observed in other patient groups 13, supporting the concept that Vericiguat treatment may result in greater improvements in vascular function in those individuals who experience the largest reductions in vascular inflammation.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic symptomatic HF (ACC/AHA Class C) and New York Heart Association (NYHA) Class II or III symptoms at the time of enrollment.
* Left ventricular ejection fraction (LVEF) of ≤45% assessed within 12 months prior to randomization by any imaging method.
* Systemic blood pressure ≥90/60 mmHg.
* Standard guideline-directed HF therapy.
* If female of reproductive potential, agrees to avoid becoming pregnant while receiving study drug and for 14 days after the last dose of study drug by complying with abstinence from heterosexual activity or use (or have her partner use) contraception during heterosexual activity.

Exclusion Criteria:

* Addition of a new disease-modifying HF pharmacotherapy or CRT-D in previous 4 weeks.
* Current or anticipated use of long-acting nitrates or nitric oxide (NO) donors including isosorbide dinitrate, isosorbide 5-mononitrate, pentaerythritol tetranitrate, nicorandil or transdermal nitroglycerin (NTG) patch, and molsidomine.
* Current or anticipated use of phosphodiesterase type 5 (PDE5) inhibitors such as vardenafil, tadalafil, and sildenafil.
* Current use or anticipated use of a soluble guanylate cyclase (sGC) stimulator such as riociguat.
* Known allergy or sensitivity to any sGC stimulator.
* Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2 or chronic dialysis.
* Patients who are pregnant or breastfeeding or plan to become pregnant or to breastfeed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josef Stehlik, M.D, M.P.H., Principal Investigator — University of Utah Health Science Center & Veterans Affairs Salt Lake City Healthcare System
Locations (2):
- United States (2):
  - University of Utah Hospital, Salt Lake City, Utah
  - Veterans Affairs Salt Lake City Health Care System (VAMC), Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vericiguat | Placebo
Started | 13 | 13
Completed | 13 | 12
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vericiguat | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [52 to 79] | 67 [59 to 71] | 67 [57 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
New York Heart Association Class II [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Classification measures the extent of heart failure. It classifies patients in 1 of 4 categories based on their limitations during physical activity. The limitations and symptoms are in regards to normal breathing and varying degrees in shortness of breath and angina pain.
  Class I is no symptoms and no limitations Class II is mild symptoms and slight limitations Class III is marked limitations in activity due to symptoms Class IV is severe limitations experiencing symptoms even while at rest
  Participants | 11 | 8 | 19
New York Heart Association Class III [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Classification measures the extent of heart failure. It classifies patients in 1 of 4 categories based on their limitations during physical activity. The limitations and symptoms are in regards to normal breathing and varying degrees in shortness of breath and angina pain.
  Class I is no symptoms and no limitations Class II is mild symptoms and slight limitations Class III is marked limitations in activity due to symptoms Class IV is severe limitations experiencing symptoms even while at rest
  Participants | 2 | 4 | 6
Systolic Blood Pressure (mmHg) [Median (Inter-Quartile Range); unit: mmHg] | 112 [106 to 126] | 99 [91 to 122] | 109 [97 to 124]
Diastolic Blood Pressure (mmHg) [Median (Inter-Quartile Range); unit: mmHg] | 75 [67 to 79] | 70 [62 to 75] | 71 [63 to 76]
Body Mass Index (Kg/m^2) [Median (Inter-Quartile Range); unit: Kg/m^2] | 29.3 [26.7 to 34.5] | 30.9 [29.6 to 34.0] | 30.8 [28.8 to 34.5]

OUTCOME MEASURES:

1. Primary Outcome: Flow-Mediated Dilation (FMD)
Description: Change in vascular function using flow-mediated vasodilation (FMD) test. FMD is quantified as the maximal change in brachial artery diameter following cuff release, expressed as a percentage increase from pre-occlusion values (%FMD).
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: % increase from pre-occlusion value
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 13 | 12
% increase from pre-occlusion value
  Baseline | 3.61 (2.36) | 3.66 (1.33)
  Week 12 | 4.22 (2.33) | 3.55 (2.72)

2. Secondary Outcome: Six-minute Walk Test (6MWT)
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 13 | 12
meters
  Baseline | 390 (155) | 398 (103)
  Week 12 | 388 (148) | 406 (97)

3. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire-12(KCCQ12)
Description: Change in Kansas City Cardiomyopathy Questionnaire-12(KCCQ12.) It is a 12-item self-administered questionnaire developed to independently measure the patient's perception of their health status, which includes heart failure symptoms, impact on physical and social function, and how their heart failure impacts their quality of life. Kansas City Cardiomyopathy Questionnaire-12(KCCQ-12) score is a 0-100 point scale with 0 being the worst status and 100 being the best possible status.
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 13 | 12
score on a scale
  Baseline | 63 (22) | 59 (20)
  Week 12 | 68 (24) | 66 (23)

4. Secondary Outcome: Visual Analogue Scale (VAS)
Description: Change in Visual Analogue Scale (VAS). Patient self-rated health status on a 0-100 point scale with endpoints labeled 'the best health you can imagine'(100) and the 'worst health you can imagine' (0).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 13 | 12
score on a scale
  Baseline | 55 (23) | 66 (21)
  Week 12 | 70 (20) | 72 (13)

5. Secondary Outcome: Inflammatory Biomarkers Serum Interleukin-18 (IL-18)
Description: Inflammation will be assessed by serum Interleukin-18 (IL-18) levels
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Vericiguat | Placebo
Number analyzed (Participants) | 13 | 12
pg/mL
  Baseline | 477 (275) | 339 (193)
  Week 12 | 461 (312) | 334 (205)

6. Secondary Outcome: Inflammatory Biomarkers Serum Interleukin-6 (IL-6)
Description: Inflammation will be assessed by serum Interleukin-6 (IL-6) levels
Time Frame: Baseline and 12 weeks
Population: At week 12, one sample in the vericiguat group could not be processed due to sample quality.
Measure: Count of Participants; unit: Participants
Groups:
- Vericiguat IL-6 <2.0 pg/mL: Vericiguat arm participants with IL-6 values <2 pg/mL
- Vericiguat IL-6 ≥2.0 pg/mL: Vericiguat arm participants with IL-6 values ≥2.0 pg/mL
- Placebo IL-6 <2.0 pg/mL: Placebo arm participants with IL-6 values <2 pg/mL
- Placebo IL-6 ≥2.0 pg/mL: Placebo arm participants with IL-6 values ≥2.0 pg/mL
Arm/Group | Vericiguat IL-6 <2.0 pg/mL | Vericiguat IL-6 ≥2.0 pg/mL | Placebo IL-6 <2.0 pg/mL | Placebo IL-6 ≥2.0 pg/mL
Number analyzed (Participants) | 13 | 13 | 12 | 12
Participants
  Baseline | 9 | 4 | 11 | 1
  Week 12: number analyzed (Participants) | 12 | 12 | 12 | 12
  Week 12 | 8 | 4 | 9 | 3

ADVERSE EVENTS:
Time Frame: Baseline to Week 12
Arm/Group | Vericiguat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 3/13 | 1/12
Other Adverse Events (participants affected / at risk) | 5/13 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat (N=13) | Placebo (N=12)
Hospitalization (Cardiac disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vericiguat (N=13) | Placebo (N=12)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 5 (5) | 6 (6)
Fatigue (General disorders) | 3 (3) | 3 (3)
New onset anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT05420012/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT05420012/ICF_001.pdf